CLINICAL TRIAL: NCT03745937
Title: A Phase 2a Randomized, Blinded, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of MEDI0382 in Overweight/Obese Subjects With Type 2 Diabetes Mellitus
Brief Title: A Study to Evaluate the Safety and Tolerability of MEDI0382 in Overweight and Obese Participants With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5670C00030
Record Dates: First submitted 2018-11-08; First posted 2018-11-19 (Actual); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MEDI0382, diabetes, obesity, overweight, type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Obesity; Overweight | interventions — cotadutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MEDI0382 Cohort 1 (Experimental): Participants will receive subcutaneous (SC) dose of MEDI0382 uptitrated weekly once daily up to 8 weeks during the up-titration period and thereafter once daily in 3-week treatment extension period (TEP).
  Interventions: Drug: MEDI0382
- Placebo Cohort 1 (Placebo Comparator): Participants will receive SC dose of placebo matched to MEDI0382 once daily up to 8 weeks during the uptitration period and thereafter once daily through 3 week TEP.
  Interventions: Drug: Placebo
- MEDI0382 Cohort 2 (Experimental): Participants will receive SC dose of MEDI0382 uptitrated weekly once daily up to 8 weeks during the up-titration period and thereafter once daily in 3-week TEP.
  Interventions: Drug: MEDI0382
- Placebo Cohort 2 (Placebo Comparator): Participants will receive SC dose of placebo matched to MEDI0382 once daily up to 8 weeks during the up-titration period and thereafter once daily through 3 week TEP.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MEDI0382 — Subcutaneous dose of MEDI0382 will be up-titrated weekly once daily up to 8 weeks during the uptitration period and thereafter once daily in 3-week TEP.
  Arms: MEDI0382 Cohort 1; MEDI0382 Cohort 2
Drug: Placebo — Subcutaneous dose of placebo matched to MEDI0382 will be administered once daily up to 8 weeks during the up-titration period and thereafter once daily through 3 week TEP.
  Arms: Placebo Cohort 1; Placebo Cohort 2

SUMMARY:
This is a Phase 2a, randomized, blinded, placebo-controlled study in up to 20 overweight or obese participants with type 2 diabetes mellitus. The participants will participate in the study for approximately 18 weeks, including screening, run-in and treatment periods and a safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18 to 74 years (inclusive) at screening.
2. Provision of signed and dated written informed consent (with the exception of consent for genetic and non-genetic research) prior to any study specific procedures.
3. Body mass index (BMI) between 27 and 35 kg/m^2 (inclusive) at screening.
4. Hemoglobin A1c (HbA1c) range of 6.5% to 8.5% (inclusive) at screening (Note: Participants may be re-tested for the HbA1c entry criterion only once.).
5. Willing and able to self-inject study drug for the duration of the study.
6. Diagnosed with type 2 diabetes mellitus with glucose control managed with metformin monotherapy where no significant dose change (increase or decrease >= 500 mg/day) has occurred in the three months prior to screening.
7. Female participants must have a negative pregnancy test at screening and randomization, and must not be lactating.
8. Female participants of childbearing potential who are sexually active with a male partner must be using at least one highly effective method of contraception from screening and up to 4 weeks after the last dose of study drug.

Exclusion Criteria:

1. History of, or any existing condition that, in the opinion of the investigator, would interfere with evaluation of the study drug, put the participant at risk, influence the participant's ability to participate or affect the interpretation of the results of the study and/or any participant unable or unwilling to follow study procedures during the run-in period.
2. Any participant who has received another study drug as part of a clinical study or a glucagon-like peptide-1 (GLP-1) analogue containing preparation within the last 30 days or 5 half-lives of the drug (whichever is longer) at the time of screening.
3. Concurrent participation in another study of any kind and repeat randomization in this study is prohibited.
4. Any participant who has received any of the following medications prior to the start of the study:

   * Herbal preparations or drugs licensed for control of body weight or appetite
   * Opiates, domperidone, metoclopramide, or other drugs known to alter gastric emptying
   * Antimicrobials within the quinolone, macrolide or azole class
   * Any change in antihypertensive medication
   * Aspirin (acetylsalicylic acid)
   * Paracetamol (acetaminophen) or paracetamol-containing preparations
   * Ascorbic acid (vitamin C) supplements
5. Severe allergy/hypersensitivity to any of the proposed study treatments, standardized meals, or excipients.
6. Symptoms of acutely decompensated blood glucose control (eg, thirst, polyuria, weight loss), a history of type 1 diabetes mellitus or diabetic ketoacidosis, or if the participant has been treated with daily SC insulin within 90 days prior to screening.
7. Acute pancreatitis, pancreatic amylase, and/or pancreatic lipase > 3 × upper limit of normal range (ULN); history of chronic pancreatitis; or serum triglyceride levels > 11 mmol/L (1000 mg/dL) at screening.
8. Significant inflammatory bowel disease, gastroparesis or other severe disease or surgery affecting the upper gastrointestinal tract (including weight-reducing surgery and procedures), which may affect gastric emptying or could affect the interpretation of safety and tolerability data.
9. Significant hepatic disease (except for nonalcoholic steatohepatitis (NASH) or non-alcoholic fatty liver disease without portal hypertension or cirrhosis) and/or participants with any of the following results at screening:

   * Aspartate transaminase (AST) >= 3 × ULN
   * Alanine transaminase (ALT) >= 3 × ULN
   * Total bilirubin (TBL) >= 2 × ULN
10. Impaired renal function defined as estimated glomerular filtration rate (GFR) < 60 mL/minute/1.73m^2 at screening.
11. Poorly controlled hypertension defined as:

    * Systolic blood pressure (BP) > 160 mm Hg
    * Diastolic BP or >= 90 mm Hg
12. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting 12-lead ECG or any abnormalities that may interfere with the interpretation of serial ECG changes.
13. Prolonged QT intervals corrected for heart rate or family history of long QT-segment at screening.
14. PR (PQ) interval prolongation, intermittent second or third-degree atrioventricular (AV) block, or AV dissociation.
15. Persistent or intermittent complete bundle branch block.
16. Unstable angina pectoris, myocardial infarction, transient ischemic attack, or stroke within 3 months prior to screening, or participants who have undergone percutaneous coronary intervention or a coronary artery bypass graft within the past 6 months or who are due to undergo these procedures at the time of screening.
17. Severe congestive heart failure.
18. Basal calcitonin level > 50 ng/L at screening or history/family history of medullary thyroid carcinoma or multiple endocrine neoplasia.
19. Hemoglobinopathy, hemolytic anemia or chronic anemia or any other condition known to interfere with the interpretation of HbA1c measurement.
20. History of neoplastic disease within 5 years prior to screening, except for adequately treated basal cell, squamous cell skin cancer, or in situ cervical cancer.
21. Any positive results for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.
22. History of substance dependence, alcohol abuse, or excessive alcohol intake. Participants who use benzodiazepines for chronic anxiety or sleep disorders may be permitted to enter the study.
23. Symptoms of depression or any other psychiatric disorder requiring treatment with medication.
24. History of severe allergy/hypersensitivity, including to any component of the investigational product formulation or other biological agent, or ongoing clinically important allergy/hypersensitivity.
25. Blood/plasma donation within 1 month of screening.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-05-28 (Actual); Study Completion 2019-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Research Site, Neuss, Germany

REFERENCES:
- See also: CSP redacted protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00030&attachmentIdentifier=d7d04e4c-35ff-4fcf-aaf5-702ceca70934&fileName=d5670c00030-csp-amendment-3-redacted.pdf&versionIdentifier=
- See also: SAP redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5670C00030&attachmentIdentifier=aa440ccc-99bd-4f76-949f-11807a0cbb85&fileName=d5670c00030-sap-ed-1-redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in Germany between 07Jan2019 and 28May2019.
Pre-assignment Details: A total of 20 participants were randomized to the study.
Groups:
- Placebo Cohort 1: Participants received subcutaneous (SC) dose of placebo matched to MEDI0382 once daily up to 8 weeks during the up-titration period and thereafter once daily through 3 week treatment extension period (TEP).
- MEDI0382 Cohort 1; MEDI0382 Cohort 2: Participants received SC dose of MEDI0382 up-titrated weekly once daily up to 8 weeks during the up-titration period and thereafter once daily in 3-week TEP.
- Placebo Cohort 2: Participants received SC dose of placebo matched to MEDI0382 once daily up to 8 weeks during the up-titration period and thereafter once daily through 3 week TEP.
Period: Overall Study
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Started | 2 | 6 | 3 | 9
Completed | 2 | 5 | 3 | 7
Not Completed | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Not-specifed | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: As-treated population included all participants who received any dose of study drug and analyzed according to the treatment they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2 | Total
Number analyzed (Participants) | 2 | 6 | 3 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.5 (3.5) | 65.3 (6.2) | 62.3 (3.5) | 67.1 (5.3) | 66.0 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 2 | 5
  Male | 2 | 5 | 1 | 7 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 6 | 3 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 2 | 6 | 3 | 9 | 20
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs) Through the End of the Up-titration Period
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Baseline (Day -1) through Day 56 (end of Up-titration period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants
  TEAEs | 2 | 6 | 3 | 8
  TESAEs | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With TEAEs and TESAEs Through the End of the Follow-up Period
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Baseline (Day-1) through 28 days post last dose (end of follow-up period; approximately up to 5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants
  TEAEs | 2 | 6 | 3 | 8
  TESAEs | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Abnormal Electrocardiograms (ECGs) Reported as TEAEs Through the End of the Up-titration Period
Description: Number of participants with abnormal ECGs reported as TEAEs are reported. Abnormal ECGs is defined as any abnormal findings in heart rate, RR interval, PR interval, QRS, QT intervals, and QTcF intervals from the primary lead of the digital 12-lead ECG.
Time Frame: Baseline (Day -1) through Day 56 (end of Up-titration period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants
  Atrial fibrillation | 0 | 0 | 0 | 1
  Supraventricular extrasystoles | 0 | 0 | 0 | 1
  Ventricular extrasystoles | 0 | 0 | 0 | 1
  Ventricular tachycardia | 1 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Abnormal ECGs Reported as TEAEs Through the End of the Follow-up Period
Description: as for outcome 3
Time Frame: Baseline (Day-1) through 28 days post last dose (end of follow-up period; approximately up to 5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants
  Atrial fibrillation | 0 | 0 | 0 | 1
  Supraventricular extrasystoles | 0 | 0 | 0 | 1
  Ventricular extrasystoles | 0 | 0 | 0 | 1
  Ventricular tachycardia | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs Through the End of the Up-titration Period
Description: Number of participants with abnormal vital signs reported as TEAEs are reported. Abnormal vital signs are defined as any abnormal finding in the vital sign parameters (blood pressure, heart rate, body temperature, and respiratory rate).
Time Frame: Baseline (Day -1) through Day 56 (end of Up-titration period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Participants With Abnormal Vital Signs Reported as TEAEs Through the End of the Follow-up Period
Description: as for outcome 5
Time Frame: Baseline (Day-1) through 28 days post last dose (end of follow-up period; approximately up to 5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 1 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Physical Examinations Reported as TEAEs Through the End of the Up-titration Period
Description: Number of participants with abnormal physical examinations reported as TEAEs are reported. Abnormal physical examinations findings are defined as any abnormal finding in the following body systems: immunologic/allergy; head, ears, eyes, nose, and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological psychiatric; dermatologic; hematologic/lymphatic; and, endocrine.
Time Frame: Baseline (Day -1) through Day 56 (end of Up-titration period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 3 | 0 | 4

8. Primary Outcome: Number of Participants With Abnormal Physical Examinations Reported as TEAEs Through the End of the Follow-up Period
Description: Number of participants with abnormal physical examinations reported as TEAEs are reported. Abnormal physical examination findings are defined as any abnormal finding in the following body systems: immunologic/allergy; head, ears, eyes, nose, and throat; respiratory; cardiovascular; gastrointestinal; musculoskeletal; neurological psychiatric; dermatologic; hematologic/lymphatic; and endocrine.
Time Frame: Baseline (Day-1) through 28 days post last dose (end of follow-up period; approximately up to 5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 3 | 0 | 4

9. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs Through the End of the Up-titration Period
Description: Number of participants with abnormal clinical laboratory parameters reported as TEAEs are reported. Abnormal clinical laboratory parameters defined as any abnormal finding during analysis of serum chemistry, hematology, and urine.
Time Frame: Baseline (Day -1) through Day 56 (end of Up-titration period)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 1 | 0 | 0

10. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Parameters Reported as TEAEs Through the End of the Follow-up Period
Description: as for outcome 9
Time Frame: Baseline (Day-1) through 28 days post last dose (end of follow-up period; approximately up to 5 months)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants | 0 | 1 | 0 | 0

11. Secondary Outcome: Area Under the Plasma Concentration Time Curve Over a Dosing Interval (AUCτ) of MEDI0382
Description: Area under the plasma concentration time curve over a dosing duration (AUCτ) of MEDI0382 is reported.
Time Frame: Pre-dose and at 1, 2, 4, 6, 8, 12 and 24 hours post dose on Days 1, 7, 14, 35, 42, 49 and 56; pre-dose on Days 22, 29, 70, 84; additional 48 and 72 hours post-dose on Day 84
Population: Pharmacokinetic (PK) population included all participants who received at least 1 dose of study drug and had at least one measurable concentration time point of MEDI0382. Here, only the participants with available data were analyzed for the specified time points.
Measure: Geometric Mean (Full Range); unit: ng.hr/mL
Groups:
- MEDI0382 (Cohort 1 + Cohort 2): Participants received SC dose of MEDI0382 up-titrated weekly once daily up to 8 weeks during the up-titration period and thereafter once daily in 3-week TEP, in both Cohorts 1 and 2.
Arm/Group | MEDI0382 (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15
ng.hr/mL
  Day 1: number analyzed (Participants) | 9
  Day 1 | 20.9 [15.9 to 29.0]
  Day 7: number analyzed (Participants) | 13
  Day 7 | 23.7 [17.2 to 41.3]
  Day 14: number analyzed (Participants) | 11
  Day 14 | 59.9 [35.8 to 101]
  Day 35: number analyzed (Participants) | 12
  Day 35 | 276 [183 to 694]
  Day 42: number analyzed (Participants) | 12
  Day 42 | 332 [247 to 735]
  Day 49: number analyzed (Participants) | 12
  Day 49 | 434 [308 to 752]
  Day 56: number analyzed (Participants) | 12
  Day 56 | 611 [343 to 2840]
  Day 84: number analyzed (Participants) | 12
  Day 84 | 661 [372 to 4740]

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of MEDI0382
Description: Maximum observed serum concentration (Cmax) of MEDI0382 is reported.
Time Frame: as for outcome 11
Population: The PK population included all participants who received at least 1 dose of study drug and had at least one measurable concentration time point of MEDI0382. Here, only the participants with available data were analyzed for the specified time points.
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15
ng/mL
  Day 1: number analyzed (Participants) | 14
  Day 1 | 1.02 [0.447 to 1.84]
  Day 7: number analyzed (Participants) | 13
  Day 7 | 1.35 [0.934 to 2.51]
  Day 14: number analyzed (Participants) | 11
  Day 14 | 3.43 [2.02 to 6.37]
  Day 35: number analyzed (Participants) | 12
  Day 35 | 15.3 [9.74 to 36.1]
  Day 42: number analyzed (Participants) | 12
  Day 42 | 17.8 [12.7 to 37.8]
  Day 49: number analyzed (Participants) | 12
  Day 49 | 24.9 [15.2 to 39.0]
  Day 56: number analyzed (Participants) | 12
  Day 56 | 32.8 [17.7 to 137]
  Day 84: number analyzed (Participants) | 12
  Day 84 | 35.3 [19.7 to 202]

13. Secondary Outcome: Time to Observed Maximum Serum Concentration (Tmax) of MEDI0382
Description: Time to observed maximum serum concentration (Tmax) of MEDI0382 is reported.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | MEDI0382 (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15
hours
  Day 1: number analyzed (Participants) | 14
  Day 1 | 6.02 [4.00 to 8.00]
  Day 7: number analyzed (Participants) | 13
  Day 7 | 6.00 [4.00 to 8.00]
  Day 14: number analyzed (Participants) | 11
  Day 14 | 6.00 [4.00 to 8.00]
  Day 35: number analyzed (Participants) | 12
  Day 35 | 6.00 [4.00 to 8.00]
  Day 42: number analyzed (Participants) | 12
  Day 42 | 6.00 [2.00 to 8.00]
  Day 49: number analyzed (Participants) | 12
  Day 49 | 6.00 [4.00 to 8.00]
  Day 56: number analyzed (Participants) | 12
  Day 56 | 6.00 [4.00 to 8.00]
  Day 84: number analyzed (Participants) | 12
  Day 84 | 6.00 [0.00 to 8.00]

14. Secondary Outcome: Trough Plasma Concentration (Ctrough) of MEDI0382
Description: Trough concentration is the lowest concentration reached by a drug before the next dose is administered. Trough plasma concentration (Ctrough) of MEDI0382 is reported.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Full Range); unit: ng/mL
Arm/Group | MEDI0382 (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15
ng/mL
  Day 1: number analyzed (Participants) | 0
  Day 7: number analyzed (Participants) | 10
  Day 7 | 0.551 [0.401 to 0.775]
  Day 14: number analyzed (Participants) | 11
  Day 14 | 1.46 [0.617 to 2.56]
  Day 22: number analyzed (Participants) | 11
  Day 22 | 2.01 [1.09 to 3.27]
  Day 29: number analyzed (Participants) | 11
  Day 29 | 4.65 [2.10 to 27.0]
  Day 35: number analyzed (Participants) | 12
  Day 35 | 6.92 [3.85 to 23.2]
  Day 42: number analyzed (Participants) | 12
  Day 42 | 8.85 [5.09 to 26.4]
  Day 49: number analyzed (Participants) | 12
  Day 49 | 11.0 [5.86 to 23.7]
  Day 56: number analyzed (Participants) | 12
  Day 56 | 16.3 [9.70 to 131]
  Day 70: number analyzed (Participants) | 11
  Day 70 | 13.6 [8.22 to 29.5]
  Day 84: number analyzed (Participants) | 12
  Day 84 | 18.8 [7.99 to 178]

15. Secondary Outcome: Observed Accumulation Ratio (Ro) of MEDI0382 Calculated Using AUC
Description: The Ro was calculated using the AUC method which account for the overall exposure measured using the Day 1 and specified time point (Day I). Ro = AUCtrough [Day I]/AUCtrough [Day 1]; where I is the specified day.
Time Frame: as for outcome 11
Population: as for outcome 12
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | MEDI0382 (Cohort 1 + Cohort 2)
Number analyzed (Participants) | 15
Ratio
  Day 1: number analyzed (Participants) | 9
  Day 1 | NA [NA to NA] — The data cannot be calculated; as for the specified time, Day I and Day 1 are same, so Ro could not be calculated.
  Day 7: number analyzed (Participants) | 8
  Day 7 | 1.25 [1.09 to 1.65]
  Day 14: number analyzed (Participants) | 6
  Day 14 | 1.40 [1.22 to 1.72]
  Day 35: number analyzed (Participants) | 7
  Day 35 | 1.01 [0.761 to 1.81]
  Day 42: number analyzed (Participants) | 7
  Day 42 | 0.857 [0.503 to 1.44]
  Day 49: number analyzed (Participants) | 7
  Day 49 | 0.904 [0.603 to 1.18]
  Day 56: number analyzed (Participants) | 8
  Day 56 | 1.16 [0.691 to 5.32]
  Day 84: number analyzed (Participants) | 8
  Day 84 | 1.30 [0.526 to 8.89]

16. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADA) to MEDI0382 Treatment
Description: Number of participants with positive ADA to MEDI0382 are reported.
Time Frame: Pre-dose (Day -2), Days 7, 14, 35, 42, 56; Day 21 of 3 week treatment extension, and 28 days post last dose (approximately 5 months)
Population: Immunogenicity population included all participants who received any dose of study drug, and had at least one serum sample for immunogenicity testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Participants
  Positive at baseline | 0 | 0 | 0 | 1
  Positive post-baseline | 0 | 3 | 0 | 4
  Positive at baseline and post-baseline | 0 | 0 | 0 | 1
  Not detected at baseline; positive post-baseline | 0 | 3 | 0 | 3
  Positive at baseline; not detected post-baseline | 0 | 0 | 0 | 1

17. Secondary Outcome: Change From Baseline in Daily (24 Hours) Average Glucose Levels Over Time as Measured by Continuous Glucose Monitoring (CGM)
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Data derived from CGM was used to calculate the average glucose level over 24-hour and 7-day periods to compare the glucose lowering efficacy of each dose level. During 14 days follow-up (Day 91), last observation carried forward (LOCF) approach was used to calculate the value.
Time Frame: Baseline (Day -1) through Day 56 (end of the up-titration period), Day 77 (end of the treatment extension period) and Day 91 (end of the follow-up period)
Population: Intent-to-treat (ITT) population included all participants who received any dose of study drug and analyzed according to their randomized treatment group. Here, only the participants with available data were analyzed for the specified time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
mg/dL
  Day 56: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 | -14.96 (16.06) | -52.04 (21.73) | -22.51 (22.41) | -34.25 (14.69)
  Day 77: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 | -10.41 (0.17) | -49.24 (25.81) | -32.54 (26.78) | -39.70 (21.85)
  Day 91: number analyzed (Participants) | 2 | 6 | 3 | 8
  Day 91 | -1.80 (25.06) | -5.71 (29.28) | 20.28 (33.40) | -13.03 (24.54)

18. Secondary Outcome: Change From Baseline in 7-day Average Glucose Levels Over Time as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Data derived from CGM was used to calculate the average glucose level over 24-hour and 7-day periods to compare the glucose lowering efficacy of each dose level.
Time Frame: Baseline (Days -7 to -1), Days 1-7, Days 8-14, Days 15-21, Days 22-28, Days 29-35, Days 36-42, Days 43-49, Days 50-56 of the Up-titration period, and Days 71-77 of end of the treatment extension period
Population: An ITT population included all participants who received any dose of study drug and analyzed according to their randomized treatment group. Here, only the participants with available data were analyzed for the specified time points.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
mg/dL
  Days 1-7: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1-7 | 37.53 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -34.64 (15.48) | -3.96 (3.30) | -26.06 (9.47)
  Days 8-14: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8-14 | 22.73 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -52.07 (19.14) | -14.44 (9.33) | -39.86 (10.44)
  Days 15-21: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15-21 | 13.83 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -44.84 (22.06) | -13.72 (18.47) | -38.10 (16.50)
  Days 22-28: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22-28 | 12.54 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -53.38 (29.90) | 5.88 (7.54) | -25.10 (33.72)
  Days 29-35: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29-35 | 16.11 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -63.28 (22.23) | 0.32 (13.60) | -40.83 (20.31)
  Days 36-42: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36-42 | 22.29 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -47.97 (24.65) | -20.03 (7.97) | -35.45 (26.96)
  Days 43-49: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43-49 | 5.69 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -48.06 (19.98) | -19.88 (29.62) | -46.84 (20.92)
  Days 50-56: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50-56 | 2.02 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -55.21 (22.32) | -19.59 (21.63) | -37.89 (18.28)
  Days 71-77: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71-77 | 21.50 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -62.66 (28.88) | -19.06 (23.43) | -40.20 (31.70)

19. Secondary Outcome: Percentage Change From Baseline in Glucose Area Under Concentration Time-curve Over 4 Hours (AUC4Hrs) During a Standardized Breakfast, Lunch, and Evening Meal Over Time as Measured by CGM
Description: Change from baseline in percentage of glucose AUC4Hrs during a standardized breakfast, lunch, and evening meal over time is reported. Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Data derived from CGM was used to calculate the average glucose level over 24-hour and 7-day periods to compare the glucose lowering efficacy of each dose level.
Time Frame: Baseline (Day -1) through Day 7 (end of Week 1), Day 56 (end of the up-titration period), and Day 77 (end of the treatment extension period)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent change in Glucose AUC4Hrs
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percent change in Glucose AUC4Hrs
  Day 7 - Breakfast: number analyzed (Participants) | 2 | 4 | 3 | 8
  Day 7 - Breakfast | -3.72 (5.73) | -27.90 (2.98) | -8.66 (6.75) | -25.85 (7.33)
  Day 56 - Breakfast: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 - Breakfast | -21.96 (13.09) | -42.22 (10.32) | -10.18 (9.18) | -32.82 (10.82)
  Day 77 - Breakfast: number analyzed (Participants) | 2 | 5 | 3 | 6
  Day 77 - Breakfast | -10.54 (6.18) | -41.52 (9.97) | -19.21 (7.20) | -32.48 (12.18)
  Day 7 - Lunch: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 - Lunch | -3.06 (23.08) | -32.55 (10.32) | 0.32 (9.00) | -15.68 (17.75)
  Day 56 - Lunch: number analyzed (Participants) | 2 | 3 | 3 | 7
  Day 56 - Lunch | -7.35 (11.46) | -33.67 (22.60) | -24.06 (10.65) | -18.30 (13.96)
  Day 77 - Lunch: number analyzed (Participants) | 2 | 3 | 3 | 7
  Day 77 - Lunch | -7.76 (20.13) | -31.10 (32.74) | -28.75 (15.12) | -21.58 (15.09)
  Day 7 - Evening Meal: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 - Evening Meal | -7.81 (17.77) | -16.14 (15.55) | -10.37 (11.55) | -22.58 (8.20)
  Day 56 - Evening Meal: number analyzed (Participants) | 2 | 5 | 2 | 7
  Day 56 - Evening Meal | -11.07 (1.26) | -35.39 (22.14) | -22.08 (13.93) | -31.44 (10.51)
  Day 77 - Evening Meal: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 - Evening Meal | -12.12 (4.61) | -26.09 (21.61) | -22.06 (14.63) | -34.18 (15.11)

20. Secondary Outcome: Change From Baseline in Coefficient of Variation (CV) in Glucose Over 7 Days as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Data derived from CGM was used to calculate the average glucose level over 24-hour and 7-day periods to compare the glucose lowering efficacy of each dose level. Change from baseline in coefficient of variation in glucose over 7 days is reported.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent of CV
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percent of CV
  Days 1 - 7: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1 - 7 | -4.48 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -0.96 (4.99) | 1.51 (3.84) | -2.41 (3.60)
  Days 8 - 14: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8 - 14 | -3.67 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.97 (4.34) | 2.26 (3.54) | -0.95 (5.62)
  Days 15 - 21: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15 - 21 | -8.86 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.65 (5.40) | -1.54 (1.05) | -4.44 (2.77)
  Days 22 - 28: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22 - 28 | -4.79 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -3.70 (6.86) | -2.49 (2.41) | -1.56 (5.23)
  Days 29 - 35: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29 - 35 | -7.92 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -5.84 (5.42) | -3.24 (1.68) | -2.52 (5.57)
  Days 36 - 42: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36 - 42 | 0.93 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -4.96 (6.54) | 1.39 (1.69) | -1.38 (4.68)
  Days 43 - 49: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43 - 49 | -3.96 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -3.68 (5.42) | 2.18 (5.40) | -1.98 (3.48)
  Days 50 - 56: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50 - 56 | -2.97 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.94 (4.61) | 4.10 (2.60) | -2.36 (3.23)
  Days 71 - 77: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71 - 77 | -4.91 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.15 (4.88) | 2.60 (2.21) | -0.82 (3.73)

21. Secondary Outcome: Change From Baseline in Percentage of Time Spent in Hyperglycemia, Normoglycemia, and Clinically Significant Hypoglycemia Over 24 Hours Time as Measured by CGM
Description: Continuous glucose monitoring is a minimally invasive device applied to the skin in the upper arm that provides a measure of interstitial glucose levels every 15 minutes. Data derived from CGM was used to calculate the average glucose level over 24-hour and 7-day periods to compare the glucose lowering efficacy of each dose level. Hyperglycemia (> 140 mg/dL), normoglycemia (70 -140 mg/dL), and clinically significant hypoglycemia (< 54 mg/dL).
Time Frame: Baseline (Day -1), Days 7, 14, 21, 28, 35, 42, 49, 56 of the up-titration period, and Day77 (end of the treatment extension period)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage of time spent
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percentage of time spent
  Day 7 - Hyperglycemia: number analyzed (Participants) | 2 | 4 | 3 | 8
  Day 7 - Hyperglycemia | -19.79 (32.41) | -39.06 (15.18) | -7.29 (14.77) | -22.66 (18.06)
  Day 14 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 - Hyperglycemia | -5.73 (12.52) | -41.67 (12.17) | -15.63 (27.14) | -25.91 (24.31)
  Day 21 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 21 - Hyperglycemia | -3.65 (8.10) | -38.50 (13.38) | 10.42 (16.04) | -22.92 (30.64)
  Day 28 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 28 - Hyperglycemia | -9.90 (18.41) | -33.54 (28.12) | 13.19 (33.09) | -21.88 (25.20)
  Day 35 - Hyperglycemia: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 35 - Hyperglycemia | -6.01 (6.84) | -51.24 (8.80) | 2.49 (25.74) | -32.30 (27.21)
  Day 42 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 - Hyperglycemia | -19.80 (7.37) | -38.33 (28.49) | -20.49 (32.81) | -36.85 (27.44)
  Day 49 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 49 - Hyperglycemia | 9.90 (19.89) | -49.79 (5.58) | -16.32 (41.07) | -42.71 (27.02)
  Day 56 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 - Hyperglycemia | -20.31 (3.68) | -50.21 (18.51) | -16.96 (26.89) | -31.40 (28.11)
  Day 77 - Hyperglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 - Hyperglycemia | -21.35 (14.00) | -46.04 (20.90) | -26.74 (30.09) | -35.27 (32.58)
  Day 7 - Normoglycemia: number analyzed (Participants) | 2 | 4 | 3 | 8
  Day 7 - Normoglycemia | 19.27 (31.67) | 39.58 (13.79) | 7.64 (15.36) | 22.66 (18.04)
  Day 14 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 - Normoglycemia | 5.21 (11.79) | 41.25 (10.25) | 13.89 (29.47) | 25.78 (24.35)
  Day 21 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 21 - Normoglycemia | 3.13 (8.84) | 39.06 (14.23) | -11.11 (16.84) | 19.53 (30.77)
  Day 28 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 28 - Normoglycemia | 9.90 (18.41) | 20.21 (18.69) | -13.54 (34.34) | 21.13 (25.07)
  Day 35 - Normoglycemia: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 35 - Normoglycemia | 5.48 (7.60) | 39.35 (10.46) | -2.14 (26.29) | 27.81 (27.30)
  Day 42 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 - Normoglycemia | 19.79 (7.37) | 34.58 (26.78) | 16.67 (37.80) | 36.72 (27.45)
  Day 49 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 49 - Normoglycemia | -10.42 (20.62) | 47.92 (5.46) | 4.86 (37.81) | 41.82 (28.31)
  Day 56 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 - Normoglycemia | 19.79 (4.42) | 40.42 (24.78) | 17.31 (27.47) | 30.51 (29.37)
  Day 77 - Normoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 - Normoglycemia | 18.75 (14.73) | 43.13 (19.72) | 21.88 (29.04) | 27.73 (36.31)
  Day 7 - Hypoglycemia: number analyzed (Participants) | 2 | 4 | 3 | 8
  Day 7 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 14 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 21 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 21 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 28 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 28 - Hypoglycemia | 0.00 (0.00) | 1.04 (2.33) | 0.00 (0.00) | 0.00 (0.00)
  Day 35 - Hypoglycemia: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 35 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 42 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 49 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 49 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 56 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 - Hypoglycemia | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Day 77 - Hypoglycemia: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 - Hypoglycemia | 0.00 (0.00) | 0.83 (1.86) | 0.00 (0.00) | 1.73 (3.73)

22. Secondary Outcome: Change From Baseline in Percentage of Time Spent in Hyperglycemia, Normoglycemia, and Clinically Significant Hypoglycemia Over 7 Days as Measured by CGM
Description: as for outcome 21
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage of time spent
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percentage of time spent
  Days 1 - 7 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1 - 7 (Hyperglycemia) | 20.70 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -32.73 (12.03) | -8.87 (5.08) | -23.38 (15.92)
  Days 8 - 14 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8 - 14 (Hyperglycemia) | 17.22 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -46.85 (16.11) | -17.00 (10.30) | -35.82 (20.15)
  Days 15 - 21 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15 - 21 (Hyperglycemia) | 19.80 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -40.52 (19.30) | -9.16 (14.98) | -33.74 (26.94)
  Days 22 - 28 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22 - 28 (Hyperglycemia) | 12.25 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -40.92 (29.12) | 6.55 (12.31) | -26.31 (25.76)
  Days 29 - 35 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29 - 35 (Hyperglycemia) | 20.10 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -51.69 (17.49) | 4.03 (15.26) | -38.19 (31.32)
  Days 36 - 42 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36 - 42 (Hyperglycemia) | 11.77 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -42.48 (25.55) | -17.21 (7.69) | -37.81 (30.52)
  Days 43 - 49 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43 - 49 (Hyperglycemia) | 9.08 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -41.92 (19.10) | -16.46 (21.74) | -44.62 (30.95)
  Days 50 - 56 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50 - 56 (Hyperglycemia) | 6.82 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -47.70 (21.30) | -18.70 (16.86) | -34.90 (27.76)
  Days 71 - 77 (Hyperglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71 - 77 (Hyperglycemia) | 18.57 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -53.98 (27.16) | -16.06 (17.53) | -40.21 (37.99)
  Days 1 - 7 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1 - 7 (Normoglycemia) | -19.94 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 32.58 (11.48) | 9.10 (5.99) | 23.34 (15.55)
  Days 8 - 14 Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8 - 14 Normoglycemia) | -16.47 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 43.41 (11.65) | 17.07 (10.85) | 33.32 (20.61)
  Days 15 - 21 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15 - 21 (Normoglycemia) | -19.20 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 40.36 (19.14) | 9.30 (15.08) | 31.82 (27.12)
  Days 22 - 28 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22 - 28 (Normoglycemia) | -12.10 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 32.09 (24.74) | -6.27 (12.58) | 22.44 (26.08)
  Days 29 - 35 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29 - 35 (Normoglycemia) | -19.49 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 42.95 (16.13) | -3.71 (15.81) | 36.13 (30.86)
  Days 36 - 42 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36 - 42 (Normoglycemia) | -11.31 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 40.62 (24.51) | 17.15 (8.75) | 37.45 (29.72)
  Days 43 - 49 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43 - 49 (Normoglycemia) | -8.63 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 40.85 (17.93) | 14.07 (19.02) | 42.81 (30.11)
  Days 50 - 56 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50 - 56 (Normoglycemia) | -6.37 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 44.10 (19.74) | 18.10 (14.94) | 33.61 (27.62)
  Days 71 - 77 (Normoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71 - 77 (Normoglycemia) | -18.27 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 46.39 (29.99) | 15.08 (17.47) | 37.93 (38.28)
  Days 1 - 7 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1 - 7 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Days 8 - 14 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8 - 14 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 1.20 (1.68) | 0.00 (0.00) | 0.28 (0.68)
  Days 15 - 21 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15 - 21 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.00 (0.00) | 0.00 (0.00) | 0.20 (0.49)
  Days 22 - 28 Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22 - 28 Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 1.09 (2.28) | 0.00 (0.00) | 0.79 (1.76)
  Days 29 - 35 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29 - 35 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.27 (0.61) | 0.00 (0.00) | 0.00 (0.00)
  Days 36 - 42 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36 - 42 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.00 (0.00) | 0.00 (0.00) | 0.00 (0.00)
  Days 43 - 49 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43 - 49 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.09 (0.20) | 0.40 (0.70) | 0.15 (0.37)
  Days 50 - 56 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50 - 56 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 0.06 (0.14) | 0.20 (0.35) | 0.15 (0.37)
  Days 71 - 77 (Hypoglycemia): number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71 - 77 (Hypoglycemia) | 0.00 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | 2.16 (3.23) | 0.15 (0.26) | 0.44 (0.59)

23. Secondary Outcome: Change From Baseline in Estimated Hemoglobin A1c (HbA1c) Based on 7-day CGM Glucose Over Time
Description: Change from baseline in estimated HbA1c based on 7-day glucose over time is reported.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percent of HbA1C
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percent of HbA1C
  Days 1 - 7: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 1 - 7 | 1.31 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.21 (0.54) | -0.14 (0.12) | -0.91 (0.33)
  Days 8 - 14: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 8 - 14 | 0.79 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.81 (0.67) | -0.50 (0.33) | -1.39 (0.36)
  Days 15 - 21: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 15 - 21 | 0.48 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.56 (0.77) | -0.48 (0.64) | -1.33 (0.58)
  Days 22 - 28: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 22 - 28 | 0.44 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.86 (1.04) | 0.21 (0.26) | -0.88 (1.18)
  Days 29 - 35: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 29 - 35 | 0.56 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.21 (0.78) | 0.01 (0.47) | -1.42 (0.71)
  Days 36 - 42: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 36 - 42 | 0.78 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.67 (0.86) | -0.70 (0.28) | -1.24 (0.94)
  Days 43 - 49: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 43 - 49 | 0.20 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.68 (0.70) | -0.69 (1.03) | -1.63 (0.73)
  Days 50 - 56: number analyzed (Participants) | 1 | 5 | 3 | 6
  Days 50 - 56 | 0.07 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -1.92 (0.78) | -0.68 (0.75) | -1.32 (0.64)
  Days 71 - 77: number analyzed (Participants) | 1 | 5 | 3 | 5
  Days 71 - 77 | 0.75 (NA) — Standard deviation is not reported as only one participant was evaluable for the specified arm. | -2.18 (1.01) | -0.66 (0.82) | -1.40 (1.10)

24. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time
Description: Change from baseline in fasting plasma glucose over time is reported. During the Day 21, and Day 28, LOCF approach was used to calculate the value.
Time Frame: as for outcome 21
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
mg/dL
  Day 7: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 | 9.0 (48.1) | -32.0 (17.7) | 13.7 (7.5) | -27.1 (12.6)
  Day 14: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 | -17.5 (31.8) | -48.0 (19.2) | -3.3 (23.9) | -33.9 (19.1)
  Day 21: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 21 | -17.5 (31.8) | -48.0 (19.2) | -3.3 (23.9) | -33.9 (19.1)
  Day 28: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 28 | -17.5 (31.8) | -48.0 (19.2) | -3.3 (23.9) | -33.9 (19.1)
  Day 35: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 35 | 28.5 (16.3) | -46.8 (25.8) | 5.7 (29.2) | -44.4 (15.8)
  Day 42: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 | 9.0 (14.1) | -42.6 (24.5) | 2.0 (27.9) | -35.1 (24.6)
  Day 49: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 49 | 23.5 (20.5) | -45.6 (23.0) | -0.3 (35.6) | -38.1 (23.7)
  Day 56: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 56 | -7.5 (37.5) | -52.8 (24.4) | -9.7 (26.4) | -31.3 (24.6)
  Day 77: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 | 1.0 (21.2) | -47.6 (34.2) | -9.7 (32.9) | -28.6 (20.5)

25. Secondary Outcome: Change From Baseline in HbA1c
Description: Change from baseline in HbA1c is reported.
Time Frame: Baseline (Day -1) through Day 77 (end of the treatment extension period)
Population: An ITT population included all participants who received any dose of study drug and analyzed according to their randomized treatment group.
Measure: Mean (Standard Deviation); unit: Percent of HbA1C
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percent of HbA1C | 0.10 (0.00) | -1.44 (0.52) | -0.40 (0.35) | -0.59 (0.74)

26. Secondary Outcome: Absolute Change From Baseline in Body Weight
Description: Absolute change from baseline in body weight is reported.
Time Frame: Baseline (Day -1) through Day 56 (end of the up-titration period) and Day 77 (end of the TEP)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Kg
  Day 56: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 56 | -0.30 (0.00) | -5.27 (3.92) | -1.70 (1.80) | -2.89 (4.15)
  Day 77: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 | -1.25 (0.64) | -6.96 (4.66) | -1.50 (1.56) | -4.56 (4.41)

27. Secondary Outcome: Percentage Change From Baseline in Body Weight
Description: Percentage change from baseline in body weight is reported.
Time Frame: Baseline (Day -1) through Day 56 (end of the up-titration period) and Day 77 (end of the TEP)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percentage change in body weight
  Day 56: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 56 | -0.33 (0.01) | -5.06 (3.16) | -1.96 (2.09) | -3.20 (4.78)
  Day 77: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 | -1.38 (0.74) | -6.88 (3.81) | -1.76 (1.79) | -5.08 (5.00)

28. Secondary Outcome: Absolute Change From Baseline in Body Weight to the End of Each Week of the Up-titration Period
Description: Absolute change from baseline in body weight to the end of each week of the up-titration period is reported.
Time Frame: Baseline (Day -1), Days 7, 14, 35, 42, 49, and 56
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Kg
  Day 7: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 | -2.05 (1.06) | -1.78 (0.86) | -0.70 (1.64) | 0.49 (4.87)
  Day 14: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 | -1.95 (0.35) | -2.72 (0.68) | -0.73 (1.10) | 0.08 (4.19)
  Day 35: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 35 | -0.60 (0.99) | -3.86 (3.24) | -0.27 (1.25) | -1.70 (4.37)
  Day 42: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 | -0.10 (0.14) | -4.40 (3.22) | -1.57 (1.50) | -2.00 (4.56)
  Day 49: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 49 | 0.10 (0.14) | -4.94 (3.63) | -1.57 (1.19) | -3.30 (5.08)
  Day 56: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 56 | -0.30 (0.00) | -5.27 (3.92) | -1.70 (1.80) | -2.89 (4.15)

29. Secondary Outcome: Percentage Change From Baseline in Body Weight to the End of Each Week of the Up-titration Period
Description: Percentage change from baseline in body weight to the end of each week of the up-titration period is reported.
Time Frame: Baseline (Day -1), Days 7, 14, 35, 42, 49, and 56
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Percentage change in body weight
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percentage change in body weight
  Day 7: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 | -2.22 (1.09) | -1.83 (0.95) | -0.77 (1.96) | 0.67 (5.69)
  Day 14: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 | -2.13 (0.32) | -2.76 (0.62) | -0.83 (1.30) | 0.22 (4.85)
  Day 35: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 35 | -0.64 (1.06) | -3.89 (2.99) | -0.27 (1.50) | -1.78 (4.95)
  Day 42: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 | -0.11 (0.15) | -4.43 (2.93) | -1.81 (1.74) | -2.09 (5.16)
  Day 49: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 49 | 0.11 (0.16) | -4.95 (3.32) | -1.82 (1.37) | -3.52 (5.67)
  Day 56: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 56 | -0.33 (0.01) | -5.06 (3.16) | -1.96 (2.09) | -3.20 (4.78)

30. Secondary Outcome: Percentage of Participants Achieving Greater Than 5% Body Weight Loss From Baseline to the End of the Treatment Extension Period
Description: Percentage of participants achieving greater than 5% body weight loss from baseline is reported.
Time Frame: Baseline (Day -1) through Day 77 (end of the treatment extension period)
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
Number analyzed (Participants) | 2 | 6 | 3 | 9
Percentage of participants
  Day 7: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 7 | 0 | 0 | 0 | 0
  Day 14: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 14 | 0 | 0 | 0 | 0
  Day 35: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 35 | 0 | 40 | 0 | 25
  Day 42: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 42 | 0 | 40 | 0 | 25
  Day 49: number analyzed (Participants) | 2 | 5 | 3 | 8
  Day 49 | 0 | 60 | 0 | 50
  Day 56: number analyzed (Participants) | 2 | 4 | 3 | 7
  Day 56 | 0 | 50 | 0 | 28.6
  Day 77: number analyzed (Participants) | 2 | 5 | 3 | 7
  Day 77 | 0 | 80 | 0 | 71.4

ADVERSE EVENTS:
Time Frame: Baseline (Day -1) through 28 days post last dose (approximately up to 5 months)
Arm/Group | Placebo Cohort 1 | MEDI0382 Cohort 1 | Placebo Cohort 2 | MEDI0382 Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/6 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/6 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 2/2 | 6/6 | 3/3 | 8/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=2) | MEDI0382 Cohort 1 (N=6) | Placebo Cohort 2 (N=3) | MEDI0382 Cohort 2 (N=9)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (8)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (4)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 2 (4) | 0 (0) | 4 (15)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 2 (4) | 1 (1)
Blood pressure diastolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appetite disorder (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT03745937/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/37/NCT03745937/SAP_001.pdf